CLINICAL TRIAL: NCT07041203
Title: Central Mechanisms and Treatment Response of Sodium Oxybate (Lumryz) in Spasmodic Dysphonia and Voice Tremor
Brief Title: Extended-release Sodium Oxybate (Lumryz) in Spasmodic Dysphonia and Voice Tremor
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kristina Simonyan (Other)
Responsible Party: Sponsor-Investigator, Kristina Simonyan, Professor of Otolaryngology-Head and Neck Surgery, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000919
Record Dates: First submitted 2025-06-04; First posted 2025-06-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Spasmodic Dysphonia; Laryngeal Dystonia; Voice Tremor
MeSH Terms: conditions — Dysphonia | interventions — Sodium Oxybate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Clinical response to sodium oxybate (Lumryz) (Experimental): Oral administration of sodium oxybate (1.5g, 2.0g, 2.5g, 3.0g)
  Interventions: Drug: sodium oxybate

INTERVENTIONS:
Drug: sodium oxybate — Oral administration of sodium oxybate (1.5g, 2.0g, 2.5g, 3.0g)
  Other Names: Lumryz

SUMMARY:
Using a comprehensive approach of clinico-behavioral testing and neuroimaging, the researchers will examine the clinical effects of the extended-release formulation of sodium oxybate on voice symptoms in spasmodic dysphonia in an open-label, proof-of-concept, dose-finding study.

DETAILED DESCRIPTION:
Spasmodic dysphonia (SD), or laryngeal dystonia, is a chronic, debilitating condition that selectively affects speech production due to involuntary spasms in the laryngeal muscles. SD often extends beyond the impairment of vocal communication, causing significant occupational disability and life-long social isolation. Treatment of SD is limited to injections of botulinum toxin into the vocal cords, however, it is often only partially effective and can have side effects. More than half of the people with SD have some relief from drinking alcohol. The previous studies showed that immediate-release sodium oxybate (an oral drug that acts similarly to alcohol) significantly relieves voice symptoms in patients with alcohol-responsive SD. In this study, we will examine the efficacy and safety of extended-release sodium oxybate formulation (Lumryz) as a longer-acting oral agent for the treatment of patients with alcohol-responsive SD.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and lifestyle considerations (see Lifestyle Considerations below) and availability for the duration of the study
3. Males and females
4. Age 21-80 years
5. Documented diagnosis of alcohol-responsive laryngeal dystonia
6. Documented positive response to immediate-release sodium oxybate (Xyrem) in prior studies
7. Willingness to adhere to the study intervention regimen

Exclusion Criteria:

1. The incapability of giving informed consent
2. Pregnancy or breastfeeding until a time when they are no longer pregnant or breastfeeding
3. Grade 2 or higher hepatic or renal dysfunction according to the NCI criteria
4. Moderate to severe congestive heart failure
5. Cognitive impairment (MoCA < 26)
6. Past or present suicidal ideations (according to C-SSRS)
7. Alcoholism or high risk for alcohol use disorder according to the NIAAA definition and DSM-5 criteria
8. Asymptomatic presentation due to botulinum toxin treatment until the time they are fully symptomatic and are at least 3 months after the last injection
9. Increased daytime sleepiness (Epworth Sleepiness Scale (ESS>10))
10. Past or present history of any neurological disorders (except for LD and co-occurring voice tremor), such as stroke, movement disorders, brain tumors, traumatic brain injury with loss of consciousness, ataxias, myopathies, myasthenia gravis, demyelinating diseases, alcoholism, drug dependence.
11. Past or present history of any psychiatric problems, such as schizophrenia, major and/or bipolar depression, or obsessive-compulsive disorder
12. Current use of medication(s) affecting the central nervous system
13. Past or present history of brain and/or laryngeal surgery
14. Presence of certain tattoos, ferromagnetic objects in their bodies (e.g., implanted stimulators, surgical clips, prosthesis, artificial heart valve, etc.) that are not MRI comparable and/or cannot be removed for the purpose of MRI study participation

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Lumryz | Through study completion, an average of 4 days
  The primary outcome will be the percent change from baseline in LD symptoms 60 min after each dose of drug intake
Efficacy of Lumryz | Through study completion, an average of 4 days
  The primary outcome will be the number of patients (N, % of total) with improved voice symptoms from baseline after each dose of the drug.

SECONDARY OUTCOMES:
Duration of treatment efficacy | Through study completion, an average of 4 days
  The secondary outcomes will be the duration (in hours) of Lumryz treatment efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided